CLINICAL TRIAL: NCT05491993
Title: Clinical Evaluation of the Sky Medical™ Rapid Diagnostic Test for Detection of SARS-CoV-2 Antigen
Brief Title: This Trial is a Clinical Performance Validation Study That Will Evaluate the Clinical Agreement of the Sky Medical™ Rapid Antigen Test Comparing the Antigen Rapid Test to RT-PCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sky Medical Supplies & Equipments, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SKYCOV001-2
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to validate the performance of the SARS-CoV-2 Antigen Test bioassay for rapid detection of infection when using a nasopharyngeal swab. A prospective randomized and blinded study to evaluate a rapid point of care bioassay for the detection of virus particles compared with the currently validated RT-PCR detection standard. Nasopharyngeal samples will be collected along with the current standard of care collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SARS-CoV-2 Antigen Rapid Test (Experimental): The same group of patients participated in two arms of the study. One arm was for obtaining data on the Rapid Antigen Test for Covid-19. The comparator arm was to obtain data from the RT-PCR.
  Interventions: Diagnostic Test: Sky Medical™ Rapid Antigen Test

INTERVENTIONS:
Diagnostic Test: Sky Medical™ Rapid Antigen Test — Rapid Antigen Diagnostic Test device performance comparative to RT-PCR.

SUMMARY:
Prospective study that will evaluate the clinical agreement of the Sky Medical™ Rapid Antigen Test compared to SARS-CoV-2 RT-PCR.

DETAILED DESCRIPTION:
Clinical performance characteristics of the Sky Medical™SARS-CoV-2 Antigen Rapid test was compared to a Reference Extracted EUA SARS-CoV-2 RT-PCR. The test kit was evaluated in the U.S in which patients were sequentially enrolled and tested. Symptomatic subjects were enrolled within six days of the onset of symptoms from a multi-site prospective clinical study. A total of 69 Nasopharyngeal samples, were tested in one (1) CLIA waived investigational site by five (5) minimally trained operators in the U.S during the 2022 COVID-19 season.

NP swab specimens collected from the patients with COVID-19 like symptoms in the U.S during the 2022 COVID-19 season and stored in BD universal transport media tube were provided by our site in the U.S. All the NP swab specimens were confirmed as positive or negative and validated with Ct value by the FDA EUA RT-PCR as a comparator method prior to the study. A total of 69 samples consisting of 39 confirmed positive nasopharyngeal (NP) swabs, 30 confirmed negative NP swab specimens were collected. The specimens were aliquoted, randomized, and blinded into sample panels that were tested by each operator, using the instructions provided by the Quick Reference Instructions (QRI).

All the study samples were randomized and assigned with a unique study subject ID by the sponsor prior to testing at the study site. The expected results of the samples were completely blinded to the operators. All the samples were tested by five (5) operators according to the Quick Reference Instructions only.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Subject is suspected case of COVID-19 by clinical criteria: a patient with acute respiratory tract infection (sudden onset of at least one of the following: cough, fever, shortness of breath, fatigue, decreased appetite, myalgia) AND with no other etiology that fully explains the clinical presentation, with or without a history of close contact with a confirmed or probable COVID-19 case in the last 14 days prior to onset of symptoms.
* Subject is an appropriate candidate for Nasopharyngeal sample collection.
* Subject is willing to provide Nasopharyngeal samples.

Exclusion Criteria:

* Individuals who present with 10 or greater days of Covid-19 Related Symptoms, (Fever, Cough, Fatigue, Decreased Appetite, Shortness of Breath, Myalgia) or post- defervescence and/or convalescence.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-01-11 (Estimated); Study Completion 2023-01-11 (Estimated)

PRIMARY OUTCOMES:
Percent Positive Agreement and Negative Percent Agreement | 90 Days
  Calculate the performance of the Rapid Antigen Test compared to PCR using swab samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sri Madireddy, PhD, Principal Investigator
Locations (1):
- American Research Labs, Lake Worth, Florida, United States